CLINICAL TRIAL: NCT06562829
Title: Application Effect of VR Combined With Lidocaine Local Infiltration Anesthesia in PICC Placement
Brief Title: The Main Content of This Study is to Use Virtual Reality Technology Combined With Local Anesthesia With Lidocaine Injection at Different Times to Reduce the Pain of PICC in School-age Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qi Yu (Other)
Responsible Party: Sponsor-Investigator, Qi Yu, Deputy chief nurse, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TJ-C20200505
Record Dates: First submitted 2024-08-12; First posted 2024-08-20 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Catheterization, Peripheral
Keywords: Catheterization pain,Virtual reality technology ,PICC

STUDY DESIGN:
Intervention Model Description: From May 2020 to May 2021, children requiring PICC were recruited by convenience sampling and divided into three groups: A, B and C. Group A was implanted with PICC under ultrasound guidance. Group B and group C all used VR intervention and used VR equipment 5 minutes before the operation began. Group B was anesthetized afterthe puncture needle was sent into the guide wire, and group C was anesthetized before the puncture needle was sent into the guide wire. The success rate of one puncture, pain, fear, compliance and catheterization time were compared among the three group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (No Intervention): Catheters were implanted according to PICC routine procedures:Sterilized skin -maximum sterile barrier-ultrasound-guided puncture insertion of guidewire -local infiltration anesthesia with 2% lidocaine -broad skin, insertion of skin expansion sheath -insertion of catheter
- Group B (Experimental): The virtual reality device used was PICO NE2, with accessories including helmet equipment , (with a field of view of about 98°, built-in Android 8.1 system, Qualcomm Snapdragon processor), and an infrared sensor (handle)and the VR headset was worn in the optimal state 5 minutes before catheterization.After preparing the vr device,Sterilized skin -maximum sterile barrier-ultrasound-guided puncture insertion of guidewire -local infiltration anesthesia with 2% lidocaine -broad skin, insertion of skin expansion sheath -insertion of catheter
  Interventions: Device: Virtual reality technology
- Group C (Experimental): The virtual reality device used was PICO NE2, with accessories including helmet equipment , (with a field of view of about 98°, built-in Android 8.1 system, Qualcomm Snapdragon processor), and an infrared sensor (handle)and the VR headset was worn in the optimal state 5 minutes before catheterization.After preparing the vr devicea and disinfecting the skin, local infiltration anesthesia was administered at the prepuncture site under ultrasound guidance using 0.5ml of 2% lidocaine. Approximately 2 minutes later, a skin puncture was performed and a guidewire was inserted. A broad incision was made to accommodate the torn vascular sheath for delivering the catheter to the predetermined length
  Interventions: Device: Virtual reality technology; Other: different timing of lidocaine injection

INTERVENTIONS:
Device: Virtual reality technology — Group B (Lidocaine injection after puncture): ①Download games in the VR headset in advance,The games last approximately 10-15 minutes. Games were selected based on children's preferences, and the VR headset was worn in the optimal state 5 minutes before catheterization.②Sterilized skin -maximum sterile barrier-ultrasound-guided puncture insertion of guidewire -local infiltration anesthesia with 2% lidocaine -broad skin, insertion of skin expansion sheath -insertion of catheter.
  Arms: Group B; Group C
Other: different timing of lidocaine injection — Group C (Lidocaine injection before puncture): Steps①was the same as in group B, After disinfecting the skin, local infiltration anesthesia was administered at the prepuncture site under ultrasound guidance using 0.5ml of 2% lidocaine. Approximately 2 minutes later, a skin puncture was performed and a guidewire was inserted. A broad incision was made to accommodate the torn vascular sheath for delivering the catheter to the predetermined length.
  Arms: Group C

SUMMARY:
We try to through the use of virtual reality technology in combination with lidocaine in different injection time to reduce the pain of PICC catheter school-age children. Using the convenience sampling method, the selection in May 2020, 2021 - may need to PICC placement of children as the research object, is divided into three groups A, B, c, group A in ultrasound guided by PICC placement; Group B and group C adopt VR intervention, and 5 min before the beginning of the next surgery using VR equipment. Group B was anesthetized after the needle was placed into the guide wire, and group C was anesthetized before the needle was placed into the guide wire.

DETAILED DESCRIPTION:
This study investigated the effect of VR combined with lidocaine local infiltration anesthesia in peripherally inserted central catheter (PICC) insertion, aiming to improve one-needle puncture success rate, reduce pain, reduce fear, improve compliance and catheterization time.

From May 2020 to May 2021, children requiring PICC were recruited by convenience sampling and divided into three groups: A, B and C. Group A was implanted with PICC under ultrasound guidance. Group B and group C all used VR intervention and used VR equipment 5 minutes before the operation began. Group B was anesthetized after the puncture needle was sent into the guide wire, and group C was anesthetized before the puncture needle was sent into the guide wire.The success rate of one puncture, pain, fear, compliance and catheterization time were compared among the three groups. A sample size and power analysis were conducted to determine the sample size required.The investigators assumed a medium effect size (f2 = 0.25) of the active VR. Using 2 tails and alpha = .05, a fixed-effect linear regression model would offer power greater than 0.80 with a total sample size of 159 children. To ensure adequate power, the investigators planned to recruit 56 participants for each group. Three groups were all operated by PICC specialist nurses, and the standard operation procedure of PICC catheterization was implemented in accordance with the infusion therapy nursing practice guidelines and implementation rules and the 2016 INS guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged between 6 and 12 years.
* Undergoing their inaugural ultrasound-guided PICC insertion in an up.
* Voluntarper limby participation and informed consent by parents or guardians.

Exclusion Criteria:

* Children with severe cardiocerebral conditionsor critical coagulopathies.
* Known lidocaine allergies.
* Severe mental illness or cognitive impairment in patients.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 174 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2021-04-17 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Success rate of one puncture | Immediately after the end of the catheterization
  The blood vessel was entered by one puncture, and there was no other operation to explore the subcutaneous vessel, pull out the needle or change the puncture site

SECONDARY OUTCOMES:
pain score | Immediately after the end of the catheterization
  Assessed using the Visual Analogue Scale ranging from "no pain" (0) to "the most severe pain" (10). A higher score indicates a greater degree of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Lijuan Feng, Study Director — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No